CLINICAL TRIAL: NCT02975921
Title: Efficacy of Povidone-Iodine Instillation Via Tunneled Pleural Catheters in Achieving Pleurodesis: A Randomized Controlled Trial
Brief Title: Betadine Pleurodesis Via Tunneled Pleural Catheters
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The site decided not to proceed with the protocol.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000020017
Record Dates: First submitted 2016-11-17; First posted 2016-11-29 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Pleural Effusion; Pleurodesis; Malignant Pleural Effusion; Pleural Effusion Due to Congestive Heart Failure; Pleural Effusion in Conditions Classified Elsewhere; Pleural Effusions, Chronic
Keywords: Pleural Effusion; Thoracentesis; Pleural Cavity; Pleurodesis; Tunneled Pleural Catheter
MeSH Terms: conditions — Pleural Effusion; Pleural Effusion, Malignant; Bronchiolitis Obliterans Syndrome | interventions — Povidone-Iodine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Malignant Effusion - Usual Care (No Intervention): Patients who had a pleural effusion secondary to a malignant etiology and subsequently underwent tunneled pleural catheter (TPC) placement and had usual care during and afterwards. Usual care is the TPC only with no intrapleural medications. They would have nursing care in the recovery area afterwards and home nursing three times weekly.
- Malignant Effusion with Pleurodesis (Experimental): Patients who had a pleural effusion secondary to a malignant etiology and subsequently underwent tunneled pleural catheter (TPC) placement and had intrapleural Povidone-Iodine administered at time of placement (100mL of 2% solution). They would have nursing care in the recovery area afterwards and home nursing three times weekly.
  Interventions: Drug: Povidone-Iodine
- Benign Effusion - Usual Care (No Intervention): Patients who had a pleural effusion secondary to a benign etiology and subsequently underwent tunneled pleural catheter (TPC) placement and had usual care during and afterwards. Usual care is the TPC only with no intrapleural medications. They would have nursing care in the recovery area afterwards and home nursing three times weekly.
- Benign Effusion with Pleurodesis (Experimental): Patients who had a pleural effusion secondary to a benign etiology and subsequently underwent tunneled pleural catheter (TPC) placement and had intrapleural Povidone-Iodine administered at time of placement (100mL of 2% solution). They would have nursing care in the recovery area afterwards and home nursing three times weekly.
  Interventions: Drug: Povidone-Iodine

INTERVENTIONS:
Drug: Povidone-Iodine — Intrapleural administration of Povidone-Iodine
  Other Names: Betadine
  Arms: Benign Effusion with Pleurodesis; Malignant Effusion with Pleurodesis

SUMMARY:
The purpose of this study is to determine whether betadine (povidone-iodine) instillation during routine indwelling Tunneled Pleural Catheter (TPC) placement is efficacious in promoting pleurodesis and thus reducing the time to TPC removal.

DETAILED DESCRIPTION:
Tunneled pleural catheter (TPC) placement is a routine clinical procedure used in the setting of recurrent pleural effusions. The most common clinical indication is malignant pleural effusion but these can be used in benign pleural effusions as well (such as those due to congestive heart failure, cirrhosis, etc). The primary benefit of TPC placement is relief of dyspnea without the need for recurrent procedures.

Despite success at relieving dyspnea, there are problems with the long-term placement of TPC's. One risk is infection which is estimated at 5%. Furthermore, each drainage kit costs approximately $100 and is often paid out-of-pocket by patients. Over time, this may create a substantial cost burden. Finally, most patients who undergo TPC placement require home drainage by visiting nurses. This is a significant resource utilization and it often requires interruption of a patient's home routines via the visitation requirements.

Occasionally, the effusion no longer reaccumulates following TPC placement. In malignant effusions, this pleurodesis (see below) occurs up to 50% of the time in malignant effusions. When pleurodesis occurs, the TPC may be removed by a simple office procedure.

Pleurodesis, or the act of inducing scarring and obliteration of the potential space between the visceral and parietal pleura where pleural effusions develop, is a different mechanism of providing relief of dyspnea. In the USA in particular, the most common agent used for pleurodesis (talc) is associated with complications such as respiratory failure and adult respiratory distress syndrome (ARDS), a life-threatening condition. Talc is also very expensive.

Povidone-Iodine, an agent used for pleurodesis in many other countries, has been shown to be highly efficacious when given via other modalities. Studies report a pleurodesis rate of 90+% with Povidone-Iodine. It also has a favorable safety record and is inexpensive.

Given all of these factors, the investigators propose a prospective study using Povidone-Iodine at the time of TPC placement to promote pleurodesis. The investigators hypothesize that pleurodesis will occur quickly and frequently, thus enabling removal of the TPC, thereby saving cost, risks of infection, all while improving patients quality of life.

The investigators plan on doing this by enrolling patients prospectively who are to undergo TPC placement as part of their standard care. These patients would be prospectively enrolled and randomized to receive either usual care (no pleurodesis) or the investigational medication (povidone-iodine) intrapleurally at time of procedure. The investigators would subdivide groups prospectively between patients who have malignant pleural effusions and those who have benign (non-malignant) pleural effusions.

Following TPC placement and medication administration (if necessary), nursing and investigative physicians would then immediately follow them in the recovery area (to monitor for any negative immediate outcomes such as hypertension, hypotension, reactions, or significant pain) and in clinic as per their usual care (starting 1-2 weeks after discharge and as long as necessary). The investigators would monitor them for the outcomes as noted elsewhere.

ELIGIBILITY:
Inclusion Criteria:

* Requiring Tunneled Catheter Placement for a Pleural Effusion

Exclusion Criteria:

* Patient with a nonexpandable lung
* Non-english speaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Time to Tunneled Pleural Catheter Removal | 0-6 months
  The time (in days) between Tunneled Pleural Catheter (TPC) placement to eventual removal within 6 months

SECONDARY OUTCOMES:
Pleurodesis Rate | 2 months
  Rate of patients who achieved successful pleurodesis within 2 months as defined as successful TPC removal with no reaccumulation of pleural effusion on subsequent imaging (usually 2-3 weeks later). Typical for usual care is 45-50%. In observational studies using povidone-iodine pleurodesis in other manners (not via TPC), a 90% pleurodesis rate was observed (which should be similar to our study with intervention).
Infection Rate | 6 months
  Any skin/site infections or empyemas (pleural based infections) noted within 6 months of TPC placement. The longer a TPC is in place, the higher the rate of infection we would expect. The expected infection rate is between 5-25% at 2 months and this should be dramatically lower in the intervention arm as most of them will have their TPCs removed within 1 week or so.
Death | 6 months
  Any deaths that occur and how long after TPC placement and the patients age at death. As patients are quite systemically ill when they receive TPCs, these comorbidities would be expected to be the primary drivers of patient mortality. Typical values seen in the literature is a mortality rate of 30-70% at 6 months. There should be essentially no difference between groups.
Mechanical Complications | 6 months
  Any mechanical complications related to the TPC itself such as catheter malfunction or accidental removal. This would be a rare complication and the expected rate will be <5%. The incidence of this will rise the longer it is in place for.
Baseline Borg Dyspnea Index | Baseline
  The Borg Dyspnea Index is a standardized, validated tool to measure a patient's dyspnea. This will be measured at baseline prior to Tunneled Pleural Catheter Placement.
Borg Dyspnea Index at 2 weeks | 2 weeks
  The Borg Dyspnea Index is a standardized, validated tool to measure a patient's dyspnea. This will be measured 2 weeks after tunneled pleural catheter placement.
Borg Dyspnea Index at 2 months | 2 months
  The Borg Dyspnea Index is a standardized, validated tool to measure a patient's dyspnea. This will be measured 2 months after tunneled pleural catheter placement.
Borg Dyspnea Index at 4 months | 4 months
  The Borg Dyspnea Index is a standardized, validated tool to measure a patient's dyspnea. This will be measured 4 months after tunneled pleural catheter placement.
Borg Dyspnea Index at 6 months | 6 months
  The Borg Dyspnea Index is a standardized, validated tool to measure a patient's dyspnea. This will be measured 6 months after tunneled pleural catheter placement.
Quality of Life Questionnaire at Baseline | Baseline
  Quality of Life will be measured via a WHOQOL-BREF questionnaire which is a standardized, validated tool to measure a patient's quality of life. This will be measured at baseline prior to the procedure.
Quality of Life Questionnaire at 2 weeks | 2 weeks
  Quality of Life will be measured via a WHOQOL-BREF questionnaire which is a standardized, validated tool to measure a patient's quality of life. This will be measured 2 weeks after TPC placement.
Quality of Life Questionnaire at 2 months | 2 months
  Quality of Life will be measured via a WHOQOL-BREF questionnaire which is a standardized, validated tool to measure a patient's quality of life. This will be measured 2 months after TPC placement.
Quality of Life Questionnaire at 4 months | 4 months
  Quality of Life will be measured via a WHOQOL-BREF questionnaire which is a standardized, validated tool to measure a patient's quality of life. This will be measured 4 months after TPC placement.
Quality of Life Questionnaire at 6 months | 6 months
  Quality of Life will be measured via a WHOQOL-BREF questionnaire which is a standardized, validated tool to measure a patient's quality of life. This will be measured 6 months after TPC placement.
Baseline Pain | Baseline
  Pain at baseline - immediately prior to procedure.
Pain 2 hours after procedure | 2 hours after procedure
  Pain at 2 hours after the procedure.
Pain 6 hours after procedure | 6 hours after procedure
  Pain at 6 hours after the procedure.
Immediate hemodynamic reactions following betadine administration | 0-6 hours after procedure
  Any severe hemodynamic fluctuations (such as severe hypotension or hypertension) noted after the procedure. The patient will monitored by nursing staff in a recovery area and any events will be noted immediately. The expected rate of this is <5%.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan T Puchalski, MD, MEd, Principal Investigator — Yale University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agarwal R, Khan A, Aggarwal AN, Gupta D. Efficacy & safety of iodopovidone pleurodesis: a systematic review & meta-analysis. Indian J Med Res. 2012 Mar;135(3):297-304. PMID 22561614
- [Background] Ahmed L, Ip H, Rao D, Patel N, Noorzad F. Talc pleurodesis through indwelling pleural catheters for malignant pleural effusions: retrospective case series of a novel clinical pathway. Chest. 2014 Dec;146(6):e190-e194. doi: 10.1378/chest.14-0394. PMID 25451360
- [Background] Hak CC, Sivakumar P, Ahmed L. Safety of indwelling pleural catheter use in patients undergoing chemotherapy: a five-year retrospective evaluation. BMC Pulm Med. 2016 Mar 11;16:41. doi: 10.1186/s12890-016-0203-7. PMID 26968653
- [Background] Light RW. Pleural effusions. Med Clin North Am. 2011 Nov;95(6):1055-70. doi: 10.1016/j.mcna.2011.08.005. Epub 2011 Sep 25. PMID 22032427
- [Background] Penz ED, Mishra EK, Davies HE, Manns BJ, Miller RF, Rahman NM. Comparing cost of indwelling pleural catheter vs talc pleurodesis for malignant pleural effusion. Chest. 2014 Oct;146(4):991-1000. doi: 10.1378/chest.13-2481. PMID 24832000
- [Background] Van Meter ME, McKee KY, Kohlwes RJ. Efficacy and safety of tunneled pleural catheters in adults with malignant pleural effusions: a systematic review. J Gen Intern Med. 2011 Jan;26(1):70-6. doi: 10.1007/s11606-010-1472-0. Epub 2010 Aug 10. PMID 20697963
- [Background] Walker S, Bibby AC, Maskell NA. Current best practice in the evaluation and management of malignant pleural effusions. Ther Adv Respir Dis. 2017 Feb;11(2):105-114. doi: 10.1177/1753465816671697. Epub 2016 Oct 24. PMID 27777372